CLINICAL TRIAL: NCT07286721
Title: The Effect of White Noise and Buzzy Use on Pain During Infant Vaccination: A Randomized Controlled Trial
Brief Title: White Noise and Buzzy for Reducing Pain During Infant Vaccination
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Burcu SELVI CALSIKAN, Assistant Professor, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/21
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Infant Pain Management
Keywords: Infant pain; White noise; Buzzy; Vaccination; Nursing
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White Noise Group (Experimental): Infants in this group will listen to white noise beginning approximately 1-2 minutes before the vaccination and continuing throughout the injection procedure. The white noise device will be placed safely within hearing distance of the infant. Pain will be assessed using the FLACC Pain Assessment Scale by a blinded observer and a parent.
  Interventions: Other: Standard Care (in control arm)
- Buzzy Device Group (Experimental): Infants in this group will receive vibration and cold stimulation using the Buzzy device. The device will be placed about 3 cm above the injection site 60 seconds before vaccination and will remain active until the procedure is completed. Pain will be assessed using the FLACC Pain Assessment Scale by a blinded observer and a parent.
  Interventions: Other: Standard Care (in control arm)
- Control Group (Experimental): Infants in this group will receive routine vaccination following standard clinical practice with no additional non-pharmacological intervention. Pain will be assessed using the FLACC Pain Assessment Scale by a blinded observer and a parent.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Other: Standard Care (in control arm) — White noise will be played 1-2 minutes before vaccination and continued throughout the procedure. The device will be placed within safe hearing distance of the infant. This auditory distraction method is intended to reduce procedural pain. No physical stimulation will be applied.
  The Buzzy device will be placed about 3 cm above the injection site 60 seconds before vaccination and kept active until the procedure ends. The device provides vibration and cold stimulation to decrease pain by activating competing sensory pathways.
  Infants in the control arm will receive routine vaccination with no additional intervention. No white noise, vibration, or cold stimulation will be used. Pain will be assessed according to standard observation procedures.

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of two non-pharmacological methods-white noise and the Buzzy device-in reducing pain experienced by infants during routine vaccination. Infants are known to feel pain, and untreated or poorly managed pain during early life may lead to negative short- and long-term outcomes. Therefore, identifying effective, safe, and easy-to-apply pain-reducing strategies is essential for improving infant comfort and supporting evidence-based nursing practices.

DETAILED DESCRIPTION:
Pain during routine vaccination is a common clinical challenge in infancy. Although short in duration, procedural pain can cause significant distress for infants and caregivers, and repeated painful experiences during early life have been associated with negative physiological, behavioral, and neurodevelopmental outcomes. Current guidelines from pediatric and neonatal organizations emphasize the importance of minimizing pain through safe, effective, and feasible strategies. Non-pharmacological methods such as white noise and vibration-cold devices (e.g., Buzzy) are increasingly recommended because they are simple, inexpensive, and easily integrated into routine clinical workflows. However, there is limited evidence comparing the effectiveness of these two methods specifically during infant vaccination.

This study is designed as a single-center, randomized controlled, experimental trial aimed at evaluating and comparing the effects of white noise and the Buzzy device on pain experienced by infants during vaccination. The study will be conducted at the Büyükçekmece Central Family Health Center in Istanbul, Türkiye, between October 2025 and October 2026. The target population includes healthy infants aged 0 to 6 months who are scheduled to receive the routine hexavalent vaccine (diphtheria, acellular pertussis, tetanus, inactivated polio, Haemophilus influenzae type B, and hepatitis B).

A total of 108 infants will be included based on a priori power analysis performed using G*Power software, assuming an alpha level of 0.05, a power of 95%, and an anticipated large effect size. To account for potential dropout or exclusions, 36 infants will be assigned to each of the three study groups: (1) White Noise Group, (2) Buzzy Device Group, and (3) Control Group. Randomization will be conducted by an independent statistician using stratified randomization based on infant age (2, 4, or 6 months) and sex to ensure balanced distribution across groups. The study will use a single-blind design in which the observer assessing pain scores is blinded to group assignment.

In the White Noise Group, infants will listen to white noise beginning approximately 1 to 2 minutes before the vaccination and continuing throughout the procedure. The device will be placed safely within hearing distance of the infant. In the Buzzy Group, the Buzzy device-providing combined vibration and cold stimulation-will be applied approximately 3 cm above the injection site starting 60 seconds before the injection and will remain active until the end of the vaccination. In the Control Group, infants will receive the standard vaccination procedure without additional intervention. All vaccinations will be performed by the same trained nurse to ensure procedural consistency. A parent will remain present for the infant's comfort and to assist in observing behavioral cues.

Pain will be evaluated using the validated FLACC Pain Assessment Scale (Face, Legs, Activity, Cry, Consolability), a widely used behavioral tool suitable for infants and young children. During the vaccination, pain scores will be independently assessed by both a blinded observer (trained research nurse) and the parent. The total FLACC score ranges from 0 (no pain) to 10 (severe pain). Higher scores indicate greater pain. Sociodemographic data for infants and parents will also be collected using a structured introductory information form developed from relevant literature.

Data analysis will be performed using SPSS software. Normality of continuous variables will be assessed using the Kolmogorov-Smirnov test. Depending on the distribution, appropriate parametric or non-parametric tests will be applied. Between-group comparisons for FLACC scores will be conducted using ANOVA or the Kruskal-Wallis test, with post hoc analyses performed where necessary. Descriptive statistics (mean, median, standard deviation, and percentages) will be used to summarize sample characteristics. A significance level of p < 0.05 will be used for all statistical tests.

The primary objective of this study is to determine whether white noise or the Buzzy device is more effective in reducing pain during infant vaccination compared with standard care. Secondary objectives include comparing the relative effectiveness of the two methods against each other and evaluating factors that may influence pain perception, such as infant age and sex. By generating evidence on the comparative effectiveness of these widely available non-pharmacological interventions, this study aims to support the development of best practices for infant pain management in primary care settings.

The findings may inform clinical guidelines, enhance nurse-led pain management strategies, and contribute to the broader adoption of evidence-based, non-pharmacological methods in pediatric care. If shown to be effective, these techniques may be recommended for routine use during infant vaccinations to improve comfort, reduce distress, and support family-centered care. The study also seeks to raise awareness among healthcare providers and caregivers regarding simple, safe, and practical ways to reduce procedural pain in infants.

ELIGIBILITY:
Inclusion Criteria

* Infants aged 2 to 6 months
* Receiving routine hexavalent vaccination
* Born at term (≥37 weeks gestation)
* Medically stable at the time of vaccination
* Parent or legal guardian able to provide written informed consent Exclusion Criteria
* Infants with neurological disorders or developmental delay
* Use of analgesic, antipyretic, or sedative medications within 24 hours prior to vaccination
* Skin conditions or contraindications at the injection site
* Hearing impairment that may affect response to white noise
* History of adverse reactions to vaccination
* Preterm infants (<37 weeks gestation)

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
FLACC Pain Score During Vaccination | Periprocedural (during vaccination)
  Pain during vaccination will be assessed using the FLACC Pain Assessment Scale (Face, Legs, Activity, Cry, Consolability). Scores range from 0 to 10, with higher scores indicating greater pain. Pain will be independently evaluated for each infant by a blinded observer and a parent.

SECONDARY OUTCOMES:
Agreement Between Parent and Observer FLACC Pain Scores | Immediately after vaccination
  The level of agreement between FLACC pain scores assessed by a blinded observer and a parent during infant vaccination will be evaluated. Inter-rater agreement will be analyzed to assess the reliability of observational pain assessment across the three study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Büyükçekmece Central Family Health Center, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations.